CLINICAL TRIAL: NCT04742296
Title: The Effects of Low-level Laser Therapy in Extensor Tendon Injuries Between Zones 5-8: A Randomized Controlled Trial
Brief Title: The Effects of Low-level Laser Therapy in Extensor Tendon Injuries Between Zones 5-8
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turkish League Against Rheumatism (Other)
Responsible Party: Principal Investigator, faruk erdogan, Principal Investigator, Turkish League Against Rheumatism
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRASD-FE-TEZ
Record Dates: First submitted 2021-01-27; First posted 2021-02-08 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Tendon Injury - Hand
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group of low level laser therapy (Active Comparator)
  Interventions: Device: low level laser therapy
- Sham group of low level laser therapy (Placebo Comparator)
  Interventions: Device: low level laser therapy

INTERVENTIONS:
Device: low level laser therapy — We will use laser light that has continuous wave mode, power of 100 mW, energy density of 7,5 joule/cm2, treatment time as 300 seconds.
  Other Names: Sham laser therapy

SUMMARY:
This study examines the rehabilitation results when low-level laser therapy is applied in zone 5-8 extensor tendon injuries. Rehabilitation results will be evaluated with both objective measurements and patient reported outcome measures. The study was planned as a double-blind, placebo-controlled, randomized, two-arm study. Participants in both treatment groups will be given exercise therapy in accordance with the early active mobilization protocol and appropriate splint will be given to be used while exercising.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Primary repair due to extensor tendon injury between Zones V-VIII
* Applying to the Hand Rehabilitation Policlinic at the end of the postoperative 1st week

Exclusion Criteria:

* Accompanying flexor tendon injury, fracture, vascular and / or nerve injury
* Active using of steroids or non-steroidal anti-inflammatory drugs
* Systemic infection or malignancy
* Pregnant or breastfeeding women
* Active wound infection
* Having a cognitive dysfunction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Change in total active motion degrees | Pre-intervention, immediately after the intervention, eighth week
  The difference of active range of motion (ROM) measurements between injured and non-injured digit(s). ROM measurement will be made with the help of a standard hand goniometer and the measured degree will be recorded.
Grip strength | Eighth week
  Grip strength measurement will be made with the Jamar dynamometer. The measured value will be recorded in kilograms.
Change in visual analog scale (VAS) score | Pre-intervention, immediately after the intervention, eighth week
  VAS is a scale used to assess pain. Minimum value of the scale is 0 and maximum is 10. Higher scores mean a worse outcome.
Change in metacarpophalangeal joint circumference | Pre-intervention, immediately after the intervention, eighth week
  It will be used to evaluate edema in the dorsum of the hand. Measurement will be made with the help of a tape measure. The measured value will be recorded in milimeters.

SECONDARY OUTCOMES:
Change in quick disabilities of arm, shoulder and hand (QuickDASH) score | Pre-intervention, immediately after the intervention, eighth week
  A scale used for measuring physical function and symptoms of upper extremities. Minimum value of the scale is 0 and maximum is 100. Higher scores mean a worse outcome.
Change in short form-36 (SF-36) scores | Pre-intervention, immediately after the intervention, eighth week
  A scale used for determining quality of life. This form evaluates the quality of life under 9 different headings. Minimum value of all headings is %0 and maximum is %100. Higher scores mean a better outcome.
Return to work | Eighth week
  The rehabilitation period required for patients to return to work

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Collocott SJF, Kelly E, Foster M, Myhr H, Wang A, Ellis RF. A randomized clinical trial comparing early active motion programs: Earlier hand function, TAM, and orthotic satisfaction with a relative motion extension program for zones V and VI extensor tendon repairs. J Hand Ther. 2020 Jan-Mar;33(1):13-24. doi: 10.1016/j.jht.2018.10.003. Epub 2019 Mar 21. PMID 30905495
- [Background] Poorpezeshk N, Ghoreishi SK, Bayat M, Pouriran R, Yavari M. Early Low-Level Laser Therapy Improves the Passive Range of Motion and Decreases Pain in Patients with Flexor Tendon Injury. Photomed Laser Surg. 2018 Oct;36(10):530-535. doi: 10.1089/pho.2018.4458. PMID 30300099